CLINICAL TRIAL: NCT07184307
Title: Intra-vesical Injection of Platelet-Rich Plasma Compared With Botox for Management of Patients With Refractory Overactive Bladder: A Comparative Randomized Study
Brief Title: Platelet-Rich Plasma Versus Botulinum Toxin for Refractory Overactive Bladder: A Randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tamer Abd El-Wahab Diab, Lecturer of Urology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD: 8-19-2026
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Overactive Bladder Syndrome; Urinary Urge Incontinence; Detrusor Overactivity
Keywords: Platelet-Rich Plasma; Botulinum Toxin Type A; Overactive Bladder; Refractory Overactive Bladder; Urinary Urgency; Urinary Frequency; Urge Urinary Incontinence; Detrusor Overactivity; Intravesical Injection; Regenerative Therapy
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either sub-urothelial platelet-rich plasma injections or intradetrusor botulinum toxin injections.
Who Masked: Outcomes Assessor
Masking Description: The study is single-blinded. The outcome assessors who evaluate bladder diaries, questionnaires, and urodynamic tests will be blinded to treatment assignment. Participants and treating physicians will be aware of the intervention due to differences in preparation and administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-Rich Plasma Injection (Experimental): Participants will receive intravesical platelet-rich plasma prepared from their own blood. Approximately 50 milliliters of venous blood will be processed with a two-step centrifugation protocol to concentrate platelets. Ten milliliters of platelet-rich plasma will be injected sub-urothelially at 20 sites (0.5 milliliters per site) in the posterior and lateral bladder walls under cystoscopic guidance with spinal or general anesthesia. A 16-French urethral catheter will be left overnight. A short oral antibiotic course will be given for three days.
  Interventions: Biological: Platelet-Rich Plasma
- Botulinum Toxin Injection (Active Comparator): Participants will receive intravesical injection of onabotulinumtoxinA. One hundred units of onabotulinumtoxinA will be reconstituted in 10 milliliters of saline and injected into the bladder detrusor muscle at 20 sites (0.5 milliliters per site), sparing the trigone, under cystoscopic guidance with spinal or general anesthesia. A 16-French urethral catheter will be left overnight. A short oral antibiotic course will be given for three days.
  Interventions: Drug: Intravesical Botulinum Toxin Injection

INTERVENTIONS:
Biological: Platelet-Rich Plasma — Autologous platelet-rich plasma prepared from approximately 50 milliliters of venous blood using a two-step centrifugation protocol. Ten milliliters of platelet-rich plasma are obtained and injected into the sub-urothelial layer of the bladder wall during cystoscopy under anesthesia.
  Arms: Platelet-Rich Plasma Injection
Drug: Intravesical Botulinum Toxin Injection — Botulinum toxin (100 units) reconstituted in 10 milliliters of saline and injected into the bladder detrusor muscle at multiple sites under cystoscopic guidance, sparing the trigone.
  Arms: Botulinum Toxin Injection

SUMMARY:
Overactive bladder is a common condition that causes sudden urges to urinate, frequent urination, night-time urination, and sometimes leakage of urine. Many people with overactive bladder improve with lifestyle changes and medicines. However, some patients do not respond to these standard treatments and continue to suffer from bothersome symptoms. This study is designed to help patients who have not improved with available medical therapy.

Two treatments will be compared in this research. The first treatment uses platelet-rich plasma. Platelet-rich plasma is made from a patient's own blood and contains growth factors that may help repair the lining of the bladder and improve bladder function. The second treatment uses botulinum toxin. Botulinum toxin is a protein that can reduce unwanted bladder contractions and is already approved for use in patients with overactive bladder who did not respond to other treatments.

The purpose of this study is to evaluate whether platelet-rich plasma injection into the bladder wall is safe, effective, and durable when compared with botulinum toxin injection into the bladder muscle. We believe that platelet-rich plasma may improve bladder health by encouraging tissue repair and reducing inflammation, while botulinum toxin may reduce bladder overactivity by blocking chemical signals that cause muscle contractions.

This study will take place at Benha University Hospital in Egypt. About 48 adult participants with overactive bladder that has not improved after at least six months of medical therapy will be enrolled. Participants will be randomly assigned to one of two groups. One group will receive platelet-rich plasma injections into the bladder lining, and the other group will receive botulinum toxin injections into the bladder muscle. The procedures will be performed under anesthesia using a cystoscope, which is a thin instrument inserted into the bladder.

Participants will be followed for one year. At several time points during follow-up, they will complete bladder symptom questionnaires, keep a voiding diary, and undergo urodynamic studies to measure bladder capacity and function. Researchers will also monitor safety by recording any side effects, such as urinary tract infections or temporary difficulty emptying the bladder.

The main goal of this study is to determine whether platelet-rich plasma can reduce symptoms of overactive bladder as effectively as botulinum toxin, with fewer side effects and longer-lasting results. If successful, platelet-rich plasma could offer a new treatment option for patients who continue to struggle with overactive bladder despite standard medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of urgency, frequency, nocturia, with or without urge urinary incontinence, lasting for at least 6 months
* Failure of standard medical treatment (antimuscarinics, beta-3 adrenergic agonists, or other appropriate therapy) for at least 6 months
* Willing and able to complete bladder diaries, questionnaires, and urodynamic testing
* Provides informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Previous intravesical biological therapy (e.g., platelet-rich plasma or botulinum toxin)
* Prior pelvic or bladder surgery that may affect bladder function
* Active urinary tract infection or sexually transmitted infection
* Vaginitis or chronic bacterial prostatitis
* Bladder or lower ureteral stones confirmed by imaging
* Bladder outlet obstruction on urodynamic study
* Bladder malignancy (mass on imaging or malignant cells on cytology)
* Use of indwelling urinary catheter
* Severe uncontrolled medical conditions (e.g., uncontrolled diabetes, advanced renal or hepatic impairment)
* Known hypersensitivity to botulinum toxin or contraindication to platelet-rich plasma preparation (e.g., coagulopathy, inability to discontinue anticoagulation safely)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in Overactive Bladder Symptom Score (OABSS) from baseline | Baseline and 6 months after intervention
  The Overactive Bladder Symptom Score (OABSS) is a patient-reported questionnaire with 4 items: daytime frequency (0-2), night-time frequency (0-3), urgency (0-5), and urge urinary incontinence (0-5). The total score ranges from 0 to 15, with higher scores indicating more severe symptoms. The outcome measure is the change in total OABSS score from baseline to follow-up.
Change in Maximum Cystometric Capacity (MCC) from baseline | Baseline and 6 months after intervention
  Maximum cystometric capacity (MCC) is measured during urodynamic testing as the bladder volume at which the patient can no longer delay urination, experiences strong desire to void, or involuntary detrusor contractions occur. Higher values indicate improved bladder storage capacity. The outcome measure is the change in MCC (in milliliters) from baseline to follow-up.

SECONDARY OUTCOMES:
Change in International Consultation on Incontinence Questionnaire-Overactive Bladder (ICIQ-OAB) score from baseline | Baseline, 3 months, 6 months, 9 months, and 12 months after intervention
  The ICIQ-OAB is a validated questionnaire assessing frequency, nocturia, urgency, and urge urinary incontinence. Each item is scored from 0 to 4, with a total score range of 0-16. Higher scores indicate worse symptoms. The outcome measure is the change in total ICIQ-OAB score from baseline to follow-up.
Incidence of urinary tract infection after intervention | Up to 12 months after intervention
  Culture-proven urinary tract infection identified during follow-up visits or patient-reported symptoms confirmed with laboratory testing. Outcome measure is the number and proportion of participants experiencing at least one urinary tract infection.
Incidence of urinary retention requiring catheterization | Up to 12 months after intervention
  Post-procedure urinary retention defined as inability to void with post-void residual volume greater than 300 milliliters, requiring temporary catheterization. Outcome measure is the number and proportion of participants who develop urinary retention.
Incidence of hematuria following intervention | Within 7 days of intervention
  Visible or microscopic hematuria documented within 7 days of the procedure. Outcome measure is the number and proportion of participants with procedure-related hematuria.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Faculty of Medicine, Department of Urology, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including baseline characteristics, outcome measures, and safety data, will be made available to other qualified researchers for secondary analyses. Personal identifiers will be removed prior to sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified IPD and supporting documents will be available beginning 12 months after publication of the primary study results and will remain available for 5 years.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal that has been approved by the Research Ethics Committee of Benha Faculty of Medicine. Requests should be submitted to the principal investigator via institutional email. Data access will be provided through secure, password-protected electronic transfer.